CLINICAL TRIAL: NCT01721096
Title: XIENCE PRIME Everolimus Eluting Coronary Stent Post Marketing Surveillance (PMS) in Japan
Brief Title: XIENCE PRIME Japan Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-398
Record Dates: First submitted 2012-09-20; First posted 2012-11-05 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-05

CONDITIONS: Angina; Coronary Occlusion; Coronary Artery Disease; Coronary Artery Stenosis; Myocardial Ischemia
Keywords: Angioplasty; Drug eluting stents; Stents; Real world
MeSH Terms: conditions — Angina Pectoris; Coronary Occlusion; Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- XIENCE PRIME - Long Length (LL): Long Lesion Arm patients (n=323) are treated by at least one Long Size stent (28, 33 and 38 mm length).There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted, and target lesion characteristics other than lesion lengths.
  Interventions: Device: XIENCE PRIME - Long Length (LL)
- XIENCE PRIME - Core Size: Core Size Arm patients (n=213) are treated with small size stent (8, 12, 15, 18 and 23 mm length). There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted, and target lesion characteristics other than lesion lengths.
  Interventions: Device: XIENCE PRIME - Core Size

INTERVENTIONS:
Device: XIENCE PRIME - Long Length (LL) — Long Length
  Groups: XIENCE PRIME - Long Length (LL)
Device: XIENCE PRIME - Core Size — Core Size
  Groups: XIENCE PRIME - Core Size

SUMMARY:
The objectives of the PMS are to observe the frequency, type, and degree of device deficiency to assure the safety of the new medical device (XIENCE PRIME) as well as to collect information on evaluation of the efficacy and safety for reevaluation.

DETAILED DESCRIPTION:
The primary objectives of the PMS are to observe the frequency, type, and degree of device deficiency to assure the safety of the new medical device (XIENCE PRIME) as well as to collect information on evaluation of the efficacy and safety for reevaluation by Pharmaceuticals and Medical Devices Agency (PMDA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic heart disease who are eligible for treatment with XIENCE PRIME Everolimus Eluting Stent
* Patient provides Informed Consent Form

Exclusion Criteria:

* If it is known at the time of index procedure that the patient is not able to return for the 8-month follow-up visit for angiogram and for the 1-year clinical follow-up, then the patient should not be registered in the PMS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only patients in Japan, who are eligible to receive treatment for coronary arteries using the XIENCE PRIME Everolimus-Eluting Stent System are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kozuma, MD, Study Chair — Teikyo University Hospital, Tokyo
Locations (1):
- Abbott Vascular Japan Co., Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 536 patients (213 in the Core Size (CS) arm and 323 in the Long Length (LL) arm) were recruited from the 25 sites between October 11, 2013 and June 30, 2013. All the patients except those terminated the surveillance have completed their follow-up at the end of the study.
Pre-assignment Details: To date, out of 536 patients, 524 (320 in LL arm and 204 in CS arm) have terminated the surveillance before completing their follow-ups
Groups:
- XIENCE PRIME - Long Length (LL): Long Lesion Arm patients (n=323) are treated by at least one Long Size stent (28, 33 and 38 mm length). There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted and target lesion characteristics other than lesion lengths.
- XIENCE PRIME - Core Size: Core Size Arm patients (n=213) are treated with small size stent (8, 12, 15, 18 and 23 mm length). There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted and target lesion characteristics other than lesion lengths.
Period: Overall Study
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Started | 323 | 213
Completed | 3 | 9
Not Completed | 320 | 204

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size | Total
Number analyzed (Participants) | 323 | 213 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (10.7) | 69.1 (10.4) | 68.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 46 | 105
  Male | 264 | 167 | 431
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 323 | 213 | 536

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Stent Thrombosis (ST)
Description: Stent thrombosis was defined by Academic Research Consortium (ARC) criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any Myocardial infarction (MI) related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis was categorized as acute (0-24 hours post stent implantation), Subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation).
Time Frame: Time Frame: Acute (0-24 hours)
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants
  Definite | 0 | 0
  Probable | 0 | 0
  Definite/Probable | 0 | 0

2. Primary Outcome: Number of Participants With Subacute Stent Thrombosis (ST)
Description: Stent thrombosis was defined by ARC criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any MI related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis was categorized as acute (0-24 hours post stent implantation), Subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation), or very late (>1 year post stent implantation).
Time Frame: Subacute (>24 hours to 30 days)
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 212
Participants
  Definite | 3 | 0
  Probable | 0 | 0
  Definite/Probable | 3 | 0

3. Primary Outcome: Number of Participants With Late Stent Thrombosis (ST)
Description: as for outcome 2
Time Frame: Late (>30 days to 1 year)
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 212
Participants
  Definite | 0 | 0
  Probable | 0 | 0
  Definite/Probable | 0 | 0

4. Primary Outcome: Total Number of Participants With Overall Stent Thrombosis
Description: as for outcome 2
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 212
Participants | 3 | 0

5. Secondary Outcome: Success Rate: Percentage of Participants With Implant Success Rate by Device
Description: Successful delivery and deployment of the first study scaffold/stent the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 50% by quantitative coronary angiography (QCA).
Time Frame: Participants will be followed for the duration of hospital stay, an average of 5 days
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
  Implant Success rate is calculated per stent base.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: Device used
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Device used) | 522 | 259
percentage of devices | 99.8 [98.9 to 100] | 99.6 [97.9 to 100]

6. Secondary Outcome: Success Rate: Percentage of Participants With Procedural Success by Lesion
Description: Achievement of final in-scaffold/stent residual stenosis of less than 50% by QCA with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (less than or equal to 7 days).
Time Frame: Participants will be followed for the duration of hospital stay, an average of 5 days
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
  Procedural Success rate is calculated per lesion base.
Measure: Number (95% Confidence Interval); unit: Percentage of Lesions
Units Other Than Participants: Lesions
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Lesions) | 402 | 241
Percentage of Lesions | 100 [99.3 to 100] | 100 [98.8 to 100]

7. Secondary Outcome: Success Rate: Percentage of Participants With Clinical Success by Patient (Per Patient Base)
Time Frame: Participants will be followed for the duration of hospital stay, an average of 5 days
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 212
percentage of participants | 100 [99.1 to 100] | 99.5 [97.4 to 100]

8. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure includes cardiac death, Target vessel MI and ischemia driven TLR
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 8 | 2

9. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure includes cardiac death, Target vessel MI and ischemia driven TLR
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 17 | 4

10. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure includes cardiac death, Target vessel MI and ischemia driven TLR
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 20 | 7

11. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure includes cardiac death, Target vessel MI and ischemia driven TLR
Time Frame: 3 years post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 23 | 7

12. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target lesion failure includes cardiac death, Target vessel MI and ischemia driven TLR
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 26 | 7

13. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 32 | 14

14. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 63 | 29

15. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 85 | 41

16. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 94 | 46

17. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 106 | 55

18. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target vessel failure includes cardiac death, MI and ischemia driven TLR; ischemia driven TVR, non TLR; ischemia driven TVR (TLR or TVR, non-TLR).
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 11 | 3

19. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 18
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 25 | 8

20. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 18
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 31 | 14

21. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 18
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 37 | 15

22. Secondary Outcome: Number of Participants With Target Vessel Failure(TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 43 | 17

23. Secondary Outcome: Number of Participants With Cardiac Death/All MI/CI-TLR (MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and ischemic driven target lesion revascularization (ID-TLR).
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 8 | 2

24. Secondary Outcome: Number of Participants With Cardiac Death/All MI/CI-TLR (MACE)
Description: as for outcome 23
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- XIENCE PRIME - Long Length (LL): Long Lesion Arm patients (n=323) are treated by at least one Long Size stent (28, 33 and 38 mm length). There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted and target lesion characteristics other than lesion lengths.
  .
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 17 | 6

25. Secondary Outcome: Number of Participants With Cardiac Death/All MI/CI-TLR (MACE)
Description: as for outcome 23
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 21 | 9

26. Secondary Outcome: Number of Participants With Cardiac Death/All MI/CI-TLR (MACE)
Description: as for outcome 23
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 26 | 9

27. Secondary Outcome: Number of Participants With Cardiac Death/All MI/CI-TLR (MACE)
Description: as for outcome 23
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 30 | 9

28. Secondary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Description: All deaths includes cardiac death, vascular death and non-cardiovascular death. Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  Non-Q wave MI: Those MIs which are not Q-wave MI
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 5 | 5

29. Secondary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Description: as for outcome 28
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 7 | 9

30. Secondary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Description: as for outcome 28
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 16 | 11

31. Secondary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Description: as for outcome 28
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 23 | 13

32. Secondary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Description: as for outcome 28
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 29 | 15

33. Secondary Outcome: Number of Participants With Cardiac Death or Myocardial Infarction (MI)
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.) Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 4 | 1

34. Secondary Outcome: Number of Participants With Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 33
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 6 | 3

35. Secondary Outcome: Number of Participants With Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 33
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 7 | 3

36. Secondary Outcome: Number of Participants With Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 33
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 10 | 3

37. Secondary Outcome: Number of Participants With Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 33
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 11 | 3

38. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI (TV-MI)
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
  TV-MI is defined as myocardial infarction attributed to target vessel myocardial infarction.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 4 | 1

39. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI (TV-MI)
Description: as for outcome 38
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 6 | 1

40. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI (TV-MI)
Description: as for outcome 38
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 6 | 1

41. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI (TV-MI)
Description: as for outcome 38
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 7 | 1

42. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI (TV-MI)
Description: as for outcome 38
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 7 | 1

43. Secondary Outcome: Number of Participants Experienced Death (Cardiac Death, Vascular Death and Non-cardiovascular Death)
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 4 | 5

44. Secondary Outcome: Number of of Participants Experienced Death (Cardiac Death, Vascular Death and Non-cardiovascular Death)
Description: as for outcome 43
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 5 | 6

45. Secondary Outcome: Number of Participants Experienced Death (Cardiac Death, Vascular Death and Non-cardiovascular Death)
Description: as for outcome 43
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 11 | 8

46. Secondary Outcome: Number of Participants Experienced Death (Cardiac Death, Vascular Death and Non-cardiovascular Death)
Description: as for outcome 43
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 16 | 11

47. Secondary Outcome: Number of Participants Experienced Death (Cardiac Death, Vascular Death and Non-cardiovascular Death)
Description: as for outcome 43
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 19 | 13

48. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 1 | 0

49. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: as for outcome 48
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 2 | 2

50. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: as for outcome 48
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 3 | 2

51. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: as for outcome 48
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 5 | 2

52. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: as for outcome 48
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 6 | 2

53. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target lesion revascularization (TLR) includes ischemia driven TLR and non-ischemia driven TLR.
  Target lesion revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 7 | 1

54. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 53
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 16 | 5

55. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 53
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 23 | 8

56. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 53
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 26 | 8

57. Secondary Outcome: Number of Participants With Target Lesion Revascularization(TLR)
Description: as for outcome 53
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 29 | 9

58. Secondary Outcome: Number of Participants With Non-Target Lesion Revascularization (Non-TLR)
Description: Non Target Lesion Revascularization (Non-TLR) is any revascularization in the target vessel for a lesion other than the target lesion.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 5 | 4

59. Secondary Outcome: Number of Participants With Non-Target Lesion Revascularization (Non-TLR)
Description: as for outcome 58
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 12 | 8

60. Secondary Outcome: Number of Participants With Non-Target Lesion Revascularization (Non-TLR)
Description: as for outcome 58
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 16 | 11

61. Secondary Outcome: Number of Participants With Non-Target Lesion Revascularization (Non-TLR)
Description: as for outcome 58
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 17 | 15

62. Secondary Outcome: Number of Participants With Non-Target Lesion Revascularization (Non-TLR)
Description: as for outcome 58
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 20 | 17

63. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: Target vessel revascularization (TLR or TVR, non-TLR) includes ischemia driven TVR (TLR or TVR non-TLR) or non-ischemia driven TVR (TLR or TVR non-TLR)
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 12 | 5

64. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR ( Non-TLR))
Description: as for outcome 63
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 28 | 13

65. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 63
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 37 | 19

66. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 63
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 41 | 23

67. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 63
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 46 | 25

68. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Any revascularization in a vessel other than the target vessel is considered as non-target vessel revascularization.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 18 | 4

69. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Any revascularization in a vessel other than the target vessel is considered as non-target vessel revascularization.
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 34 | 9

70. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Any revascularization in a vessel other than the target vessel is considered as non-target vessel revascularization.
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 43 | 15

71. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Any revascularization in a vessel other than the target vessel is considered as non-target vessel revascularization.
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 50 | 19

72. Secondary Outcome: Number of Participants With Non-Target Vessel Revascularization (Non-TVR)
Description: Any revascularization in a vessel other than the target vessel is considered as non-target vessel revascularization.
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 57 | 25

73. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven and non-ischemia driven revascularization.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 28 | 9

74. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven and non-ischemia driven revascularization.
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 57 | 22

75. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven and non-ischemia driven revascularization.
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 72 | 33

76. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven and non-ischemia driven revascularization.
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 77 | 37

77. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven and non-ischemia driven revascularization.
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 87 | 45

78. Secondary Outcome: Number of Participants Experienced Bleeding
Description: Bleeding complications will be defined according to the GUSTO (Global Use of Strategies to Open Occluded Coronary Arteries) classification of severe, moderate, and mild bleeding events.
  Severe or life-threatening: Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention Moderate: Bleeding that requires blood transfusion but does not result in hemodynamic compromise Mild: Bleeding that does not meet criteria for either moderate or severe bleeding
Time Frame: 8 months post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 0 | 1

79. Secondary Outcome: Number of Participants Experienced Bleeding
Description: as for outcome 78
Time Frame: 1 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 0 | 2

80. Secondary Outcome: Number of Participants Experienced Bleeding
Description: as for outcome 78
Time Frame: 2 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 0 | 4

81. Secondary Outcome: Number of Participants Experienced Bleeding
Description: as for outcome 78
Time Frame: 3 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 1 | 4

82. Secondary Outcome: Number of Participants Experienced Bleeding
Description: as for outcome 78
Time Frame: 4 year post index procedure
Population: The number of participants analyzed excludes subjects who were lost-to-follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Participants | 1 | 4

83. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: The value calculated as 100 * (1 - minimum lumen diameter/reference vessel diameter) (MLD/RVD) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of DS
Units Other Than Participants: Number of lesion analyzed
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Number of lesion analyzed) | 377 | 245
percentage of DS | 73.96 (17.73) | 70.27 (15.13)

84. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: The value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: Post procedure
Measure: Mean (Standard Deviation); unit: percentage of DS
Units Other Than Participants: Number of lesion analyzed
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Number of lesion analyzed) | 375 | 245
percentage of DS | 25.94 (11.76) | 23.58 (10.79)

85. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: The value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: 8 months post index procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: percentage of DS
Units Other Than Participants: Number of lesion analyzed
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 237 | 154
Number analyzed (Number of lesion analyzed) | 275 | 175
percentage of DS | 29.17 (15.50) | 25.12 (12.88)

86. Secondary Outcome: Acute Gain: In-stent, In-segment
Description: The difference between post- and pre-procedural MLD.
Time Frame: 8 months post index procedure
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Lesions) | 375 | 244
mm
  Stent | 1.81 (0.56) | 1.81 (0.53)
  Segment | 1.42 (0.62) | 1.40 (0.61)

87. Secondary Outcome: Net Gain: In-stent, In-segment
Description: Late procedural outcome is influenced by both the acute gain provided by the intervention (pre to post) and the subsequent late loss that occurs after the intervention (post to follow-up).The net gain is thus the sum of the offsetting effects of acute gain and late loss (net gain = acute gain - late loss).
Time Frame: 8 months post index procedure
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Lesions) | 273 | 174
mm
  Stent | 1.53 (0.66) | 1.68 (0.58)
  Segment | 1.31 (0.67) | 1.34 (0.64)

88. Secondary Outcome: Late Loss(LL): In-stent, In-segment, Proximal, and Distal
Description: Late loss is calculated as MLD post procedure - MLD at follow-up.
Time Frame: 8 months post index procedure
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | XIENCE PRIME - Long Length (LL) | XIENCE PRIME - Core Size
Number analyzed (Participants) | 323 | 213
Number analyzed (Lesions) | 273 | 175
mm
  Stent | 0.27 (0.41) | 0.15 (0.29)
  Proximal | 0.13 (0.44) | 0.08 (0.40)
  Distal | -0.04 (0.36) | 0.03 (0.35)
  Segment | 0.12 (0.50) | 0.06 (0.45)

ADVERSE EVENTS:
Time Frame: 4 years
Description: This Surveillance is conducted per the Ministerial Ordinance on Good PMS Practice for Medical Devices to measure the frequency&status of adverse device effects&AEs in order to assure the safety of the new medical device to be evaluated for repeat review by PMDA. PMDA has requested for a combined AE for follow up period, as the difference between both the groups are just based on length of the device,which does not signify a change in the technology but the same technology applies.
Groups:
- XIENCE PRIME - Long Length (LL) and Core Size (CS): The study has 2 arms depending upon the size of stent used for the treatment: Long Lesion Arm patients (n=323) are treated by at least one Long Size stent (28, 33 and 38 mm length), whereas Core Size Arm patients (n=213) are treated with small size stent (8, 12, 15, 18 and 23 mm length). There are no significant difference between both the groups with respect to patient background, ischemic status, risk factors and medical history, numbers of target lesions and the lesion types, target lesion treatment, number of stents implanted and target lesion characteristics other than lesion lengths.
Arm/Group | XIENCE PRIME - Long Length (LL) and Core Size (CS)
All-Cause Mortality (participants affected / at risk) | 47/536
Serious Adverse Events (participants affected / at risk) | 221/536
Other Adverse Events (participants affected / at risk) | 254/536
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE PRIME - Long Length (LL) and Core Size (CS) (N=536)
Anemia (Blood and lymphatic system disorders) | 3
Acute heart failure (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 5
Angina pectoris (Cardiac disorders) | 48
Angina unstable (Cardiac disorders) | 10
Angiopathy (Cardiac disorders) | 12
Aortic aneurysm (Cardiac disorders) | 2
Aortic dissection (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardio respiration (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Chronic heart failure (Cardiac disorders) | 7
Complete atrioventricular block (Cardiac disorders) | 1
Congestive heart failure (Cardiac disorders) | 3
Contractile pericarditis (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 47
Heart failure (Cardiac disorders) | 23
Intermittent claudication (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischemia (Cardiac disorders) | 6
Peripheral arterial obstructive disease (Cardiac disorders) | 11
Peripheral ischemia (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Second degree atrioventricular block (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 2
Supraventricular arrhythmia (Cardiac disorders) | 5
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular extrasystole (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Dizziness, vertigo (Ear and labyrinth disorders) | 1
Diabetic retinopathy (Eye disorders) | 2
Macular hole (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Atrophic gastritis (Gastrointestinal disorders) | 1
Colon Bleeding (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 5
Colorectal polyp (Gastrointestinal disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Ischemic colitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 47
Thrombosis in device (General disorders) | 3
Acute cholangitis (Hepatobiliary disorders) | 1
Acute cholecystitis (Hepatobiliary disorders) | 3
Bile duct stones (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Liver cirrhosis (Hepatobiliary disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Acute pyelonephritis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Discitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lymph node tuberculosis (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pyelonephritis (Infections and infestations) | 4
Pyoderma (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Sepsis shock (Infections and infestations) | 1
Urinary tract Infection (Infections and infestations) | 1
Cerebral contusion (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 31
Femoral fracture (Injury, poisoning and procedural complications) | 1
Graft vascular occlusion (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 2
Ligament tear (Injury, poisoning and procedural complications) | 1
Shunt obstruction (Injury, poisoning and procedural complications) | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Exercise test abnormal (Investigations) | 1
Motor test abnormality (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Crystalline joint disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral stenosis (Musculoskeletal and connective tissue disorders) | 1
Intramuscular Bleeding (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of the liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of the tongue, stage unknown (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal sigmoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Recurrent liver malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Altered state of consciousness (Nervous system disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Cerebellar infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 5
Dementia with Lewy bodies (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 2
Floating dizziness (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Lacunar infarct (Nervous system disorders) | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Chronic renal failure (Renal and urinary disorders) | 1
Kidney failure (Renal and urinary disorders) | 2
Renal dysfunction (Renal and urinary disorders) | 4
Prostatitis (Reproductive system and breast disorders) | 1
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Medical device related thrombosis (Surgical and medical procedures) | 3
Medical equipment blockage (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 4
Peripheral ischemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE PRIME - Long Length (LL) and Core Size (CS) (N=536)
Angina pectoris (Cardiac disorders) | 58
Coronary artery stenosis (Cardiac disorders) | 54
Acute myocardial infarction (Cardiac disorders) | 5
Unstable angina (Cardiac disorders) | 13
Aortic valve stenosis (Cardiac disorders) | 2
Supra ventricular arrhythmia (Cardiac disorders) | 7
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Complete atrioventricular block (Cardiac disorders) | 1
Second degree atrioventricular block (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 23
Cardio respiration (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary embolism (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischemia (Cardiac disorders) | 10
Contractile pericarditis (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular extrasystole (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Coronary dissection (Cardiac disorders) | 4
Cardiac puncture (Cardiac disorders) | 2
Coronary artery no re flow phenomenon (Cardiac disorders) | 1
Angiopathy (Cardiac disorders) | 17
Aortic aneurysm (Cardiac disorders) | 2
Aortic dissection (Cardiac disorders) | 1
Intermittent claudication (Cardiac disorders) | 1
Peripheral ischemia (Cardiac disorders) | 1
Peripheral arterial obstructive disease (Cardiac disorders) | 11
Reperfusion injury (Cardiac disorders) | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Nose bleeding (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Ischemic colitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 5
Atrophic gastritis (Gastrointestinal disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Colorectal polyp (Gastrointestinal disorders) | 1
Colon bleeding (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Acute cholecystitis (Hepatobiliary disorders) | 3
Liver cirrhosis (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Lumbar spinal canal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intramuscular hemorrhage (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Crystalline joint disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral stenosis (Musculoskeletal and connective tissue disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Renal dysfunction (Renal and urinary disorders) | 4
Prostatitis (Reproductive system and breast disorders) | 1
Asthenia (General disorders) | 1
Medical device related thrombosis (Surgical and medical procedures) | 3
Medical device obstruction (Surgical and medical procedures) | 1
Increased myocardial enzyme (Investigations) | 1
Motor test abnormality (Investigations) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Femoral fracture (Injury, poisoning and procedural complications) | 1
Shunt obstruction (Injury, poisoning and procedural complications) | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Graft vascular occlusion (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Cerebral contusion (Injury, poisoning and procedural complications) | 1
Coronary restenosis (Injury, poisoning and procedural complications) | 38
Ligament injury (Injury, poisoning and procedural complications) | 2
Ligament tear (Injury, poisoning and procedural complications) | 1
Can not pass target lesion (General disorders) | 2
Balloon rupture (Injury, poisoning and procedural complications) | 1
Tearing (Product Issues) | 1
Stent damaged / deformed after indwelling-others (Product Issues) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lymph node tuberculosis (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pyelonephritis (Infections and infestations) | 4
Pyoderma (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Abdominal segment abscess (Infections and infestations) | 1
Disc flame (Infections and infestations) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Liver malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of the tongue, stage unknown (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anemia (Blood and lymphatic system disorders) | 3
Drug hypersensitivity (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Marasmus (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Dizziness, vertigo (Ear and labyrinth disorders) | 1
Diabetic retinopathy (Eye disorders) | 2
Macular hole (Eye disorders) | 1
State of consciousness transformation (Nervous system disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Carotid stenosis (Nervous system disorders) | 2
Cerebellar infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 5
Diabetic neuropathy (Nervous system disorders) | 1
Floating dizziness (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoglycemia coma (Metabolism and nutrition disorders) | 1
Subarachnoid hemorrhage (Nervous system disorders) | 1
Transient ischemic attack (Nervous system disorders) | 1
Lacunar infarct (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 2
Lewy body dementia (Nervous system disorders) | 1
Acute heart failure (Cardiac disorders) | 1
Chronic heart failure (Cardiac disorders) | 7
Congestive heart failure (Cardiac disorders) | 3
Acute cholangitis (Hepatobiliary disorders) | 1
Acute pyelonephritis (Infections and infestations) | 1
Rectal sigmoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Chronic renal failure (Renal and urinary disorders) | 1
Kidney failure (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days